CLINICAL TRIAL: NCT02249728
Title: A Phase I , Open-Label Study to Evaluate the Absorption, Metabolism and Excretion of [14C]-PBT2 and to Estimate the Absolute Bioavailability of PBT2 in Healthy Male Subjects
Brief Title: Absorption, Metabolism and Excretion Study of [14C]PBT2 and Absolute Bioavailability of PBT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prana Biotechnology Limited (Industry)
Responsible Party: Sponsor
Organization: Pranabio (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBT2-102; 2014-000389-24 (EudraCT Number)
Record Dates: First submitted 2014-07-30; First posted 2014-09-26 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absolute Bioavailability (Experimental): IV PBT2 microtracer and oral PBT2 single dose
  Interventions: Drug: IV PBT2 microtracer and oral PBT2 single dose
- Radiolabelled AME (Experimental): oral 14C PBT2
  Interventions: Drug: oral 14C-PBT2

INTERVENTIONS:
Drug: IV PBT2 microtracer and oral PBT2 single dose
  Arms: Absolute Bioavailability
Drug: oral 14C-PBT2
  Arms: Radiolabelled AME

SUMMARY:
The purpose of the study is to investigate how the test drug, PBT2, is taken up, broken down and removed from the body when given as an oral capsule, a radiolabelled oral suspension and a radiolabelled intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Body mass index of 18.0 to 35.0 kg/m2

Exclusion Criteria:

* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of cardiovascular, renal, hepatic, chronic respiratory or GI disease as judged by the investigator

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Herd, PhD, Study Director — Prana Biotechnology Ltd
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled into one study site in the United Kingdom.
Groups:
- All Study Participants: In Part One (Absolute Bioavailability), a single dose of oral PBT2 250 mg capsule administered followed by IV PBT2 microtracer. Participants then proceed into Part Two.
  In Part Two (Radiolabelled AME), a single dose of oral PBT2 250mg 14C suspension administered
Period: Part One (4 Days)
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0
Period: Part Two (up to 6 Days)
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: In Part One (Absolute Bioavailability), a single dose of oral PBT2 250 mg capsule administered followed by IV PBT2 microtracer. Following completion of Part One, participants crossed over into Part Two (Radiolabelled AME), where a single dose of oral PBT2 250 mg 14C suspension was administered.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.55 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability of PBT2 (F%)
Description: Absolute bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose, computed as AUC(oral)/AUC(IV), with range from 0% (no drug) to 100% (all of the administered drug).
Time Frame: 0 to 72 hours post oral dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: percentage of absolute bioavailability
Groups:
- Part One Absolute Bioavailability: In Part One (Absolute Bioavailability), a single dose of oral PBT2 250 mg capsule administered followed by IV PBT2 microtracer. Participants then proceed into Part Two.
  In Part Two (Radiolabelled AME), a single dose of oral PBT2 250mg 14C suspension administered
Arm/Group | Part One Absolute Bioavailability
Number analyzed (Participants) | 6
percentage of absolute bioavailability | 15.936 (28.2)

2. Primary Outcome: Mass Balance
Description: Amount excreted as a percentage of the administered dose (%Ae)
Time Frame: 168 h (7 days) post dose
Population: PK Population
Measure: Geometric Mean (Standard Deviation); unit: percentage of administered dose
Groups:
- Part Two Radiolabelled AME: In Part One (Absolute Bioavailability), a single dose of oral PBT2 250 mg capsule administered followed by IV PBT2 microtracer. Participants then proceed into Part Two.
  In Part Two (Radiolabelled AME), a single dose of oral PBT2 250mg 14C suspension administered
Arm/Group | Part Two Radiolabelled AME
Number analyzed (Participants) | 5
percentage of administered dose | 98.65 (1.28)

3. Secondary Outcome: IV PK Profile of [14C]-PBT2 and Total Radioactivity as Assessed by AUC(0 Last)
Description: Area under the plasma concentration vs time curve from time 0h to the last time point of IV [14C]-PBT2 .
Time Frame: 0 to 72 h post oral dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Arm/Group | Part Two Radiolabelled AME
Number analyzed (Participants) | 6
ng*hr/ml | 3.40 (28.8)

4. Secondary Outcome: Oral PK Profile of PBT2 as Assessed by AUC(0-last)
Description: Area under the plasma concentration vs time curve from time 0h to the last time point of oral PBT2 .
Time Frame: 72 h post oral dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Arm/Group | Part One Absolute Bioavailability
Number analyzed (Participants) | 6
ng*hr/ml | 1330 (51.2)

5. Secondary Outcome: Safety and Tolerability of PBT2
Description: As assessed by the number of participants with adverse events
Time Frame: 72 h post oral dose
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
participants | 1

6. Secondary Outcome: Ratio of Whole Blood, Plasma [14C] PBT2 at 24 Hours
Description: Ratio of whole blood, plasma [14C] PBT2 at 24 hours
Time Frame: 0 to 24 hours
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio [14C] PBT2
Arm/Group | Part Two Radiolabelled AME
Number analyzed (Participants) | 6
ratio [14C] PBT2 | 0.488 (5.1)

7. Secondary Outcome: Oral PK Profile of [14C]-PBT2 as Assessed by AUC(0-last)
Description: area under the plasma concentration vs time curve to the last timepoint
Time Frame: 0 to 72 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part Two Radiolabelle AME: In Part One (Absolute Bioavailability), a single dose of oral PBT2 250 mg capsule administered followed by IV PBT2 microtracer. Participants then proceed into Part Two.
  In Part Two (Radiolabelled AME), a single dose of oral PBT2 250mg 14C suspension administered
Arm/Group | Part Two Radiolabelle AME
Number analyzed (Participants) | 6
ng*hr/mL | 1660 (48.3)

ADVERSE EVENTS:
Time Frame: Reported AEs from dosing in Part 1 to the end of the study (Day 15 to 20).
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=6)
Mild Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less